CLINICAL TRIAL: NCT00803179
Title: Growth Hormone Therapy for Wasting in Cystic Fibrosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor enrollment, patients were lost to follow up
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 900005
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2013-01-15 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis
Keywords: CF
MeSH Terms: conditions — Cystic Fibrosis | interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Growth Hormone Therapy (Experimental): Nutropin Aqueous (AQ):
  Initiation treatment for adult males is 0.2mg/d and for women 0.4mg/d
  Interventions: Drug: Nutropin AQ

INTERVENTIONS:
Drug: Nutropin AQ — Based on recommendations from the 2007 GH Deficiency Consensus Workshop on adult GH deficiency, the recommended initiation of treatment for adult males is 0.2mg/d and for women 0.4mg/d, with a titration upwards based on insulin-like growth factor (IGF-1) (product of GH stimulation at target tissues) levels and patient response. IGF-1 will be monitored at the 3,4,5 and 11 month intervals. For subjects under the age of 25 with an open epiphysis of the hand and/or wrist we will treat with the dose of 0.3mg/kg/week. Subjects will be on growth hormone for 8 months with a baseline visit prior to initiation of therapy and a 3 month follow-up visit after stopping therapy.
  Other Names: Growth Hormone (GH)

SUMMARY:
Our hypothesis is that Growth Hormone (GH) will not only target the peripheral tissue to stimulate weight and muscle growth which will maximize nutritional potential and improve overall quality of life. We theorize that this will occur through a multitude of factors: increased appetite, more constructive utilization of caloric intake and decreased catabolic signaling. The first aim will address changes in weight and lean body mass following the institution of GH therapy in adults with Cystic Fibrosis (CF) related wasting. The second aim will measure impact on quality of life of these individuals. Additionally, the third aim will monitor effects of GH therapy on diabetes and insulin sensitivity. Finally, the fourth aim will observe changes in the subjects underlying diagnosis of CF, specifically lung function, muscle strength and inflammatory state.

DETAILED DESCRIPTION:
The following is a more detailed description of the aims listed above:

Specific Aim 1: Measure change in weight in adults with CF related wasting following GH therapy.

1.1) Monitor weight gained or loss from baseline. 1.2) Assess changes in fat free mass from baseline by bioelectrical impedence analysis.

Specific Aim 2: Evaluate overall quality of life (QOL) in adults with CF related wasting treated with GH therapy.

2.1) Perform CF disease-specific and general QOL analysis via CF QOL questionnaires.

2.2) Monitor compliance with therapy via subject report.

Specific Aim 3: Monitor impact of GH therapy in relation to CF related diabetes onset or control.

3.1) Measure impact on insulin sensitivity in non-diabetes subjects 3.2) Observe change in exogenous insulin requirements and glycemic control in subjects with diabetes.

Specific Aim 4: Quantify impact of anabolic therapy on manifestations of underlying diagnosis associated with CF.

4.1) Observe changes in lung function from baseline during GH therapy. 4.2) Determine changes in overall muscle strength via hand grip and six minute walk.

4.3) Evaluate changes in serum markers.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Age > 18 years
* Cystic fibrosis, diagnosed by either sweat chloride or genetic testing
* Less than 92% ideal body weight based on body mass index (BMI) of 22 for women and 23 for men
* Moderate or better pulmonary function (Forced Expiratory Volume (FEV1) >40% of predicted).
* Agree to use an effective method of birth control to prevent pregnancy during the research study.

Women should not nurse (breast feed) a baby while on this study because Nutropin AQ may enter breast milk and possibly harm the child.

Exclusion Criteria:

* Pregnancy (positive pregnancy test) prior enrollment in the study
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial
* Pediatric patients
* Active neoplasm
* History of organ transplantation
* Prader Willi Syndrome who are severely obese or have severe respiratory impairment
* Patients with hepatic impairment resulting in abnormal coagulation studies (>1.5 times normal reference range)
* Poorly controlled diabetes as determined by a Hemoglobin A1c greater than or equal to 9.0%.
* Individuals with electrocardiogram abnormality or cardiac pacing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stalvey, MD, Principal Investigator — Unversity of Massachusetts Medical School
Locations (1):
- Umms/Ummhc, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Thaker V, Carter B, Putman M. Recombinant growth hormone therapy for cystic fibrosis in children and young adults. Cochrane Database Syst Rev. 2021 Aug 23;8(8):CD008901. doi: 10.1002/14651858.CD008901.pub5. PMID 34424546

RESULTS

PARTICIPANT FLOW:
Groups:
- Growth Hormone Therapy: Nutropin AQ:
  Initiation treatment for adult males is 0.2mg/d and for women 0.4mg/d
Period: Overall Study
Arm/Group | Growth Hormone Therapy
Started | 5
Completed | 2
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Growth Hormone Therapy
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Measure Change in Weight in Adults With Cystic Fibrosis (CF) Related Wasting Following Growth Hormone (GH) Therapy
Time Frame: 14 months
Population: The study was stopped prematurely due to lack of enrollment and dropout. There was not sufficient number of individuals completing the study to perform an analysis.
Arm/Group | Growth Hormone Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Evaluate Overall Quality of Life (QOL) in Adults With CF Related Wasting Treated With GH Therapy
Time Frame: 14 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Growth Hormone Therapy
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes